CLINICAL TRIAL: NCT03055455
Title: Neuroimaging and Neuromonitoring in Critically Ill Children With Sepsis
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 16-012645
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sepsis: Children with severe sepsis or septic shock
  Interventions: Diagnostic Test: MR imaging

INTERVENTIONS:
Diagnostic Test: MR imaging — Conventional structural imaging will be combined with advanced neuroimaging modalities to evaluate integrity of white matter tracts, regional brain perfusion, and the 3-dimensional volume of specific brain structures.

SUMMARY:
In critically ill children with severe sepsis, neurophysiologic derangements often proceed undetected and can lead to irreversible brain injury causing neurocognitive and behavioral deficits. The etiology of these impairments is unclear, however, it is likely that some of this neural injury is preventable. The overarching goal for this study is to show that acute acquired structural and microstructural brain injury occurs in critically ill children with severe sepsis, and that this injury is related to neuropsychological deficits and impaired cerebral autoregulation (CAR). Subjects will complete Magnetic resonance (MR) imaging within 2-10 days of recognition of their severe sepsis. Subjects will undergo serial interrogation of CAR for up to 10 days. CAR will be determined by the correlation of arterial blood pressure with middle cerebral artery flow velocity measured by transcranial doppler ultrasonography and cerebral oximetry derived from near-infrared spectroscopy. Subjects will also participate in a neuropsychological evaluation 6 months after enrollment to evaluate multiple domains of behavior and cognition.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the Children's Hospital of Philadelphia (CHOP) pediatric intensive care unit (PICU)
* Males or females ages ≥ 3.5 years and ≤ 18 years on day of sepsis recognition
* Meet published consensus criteria for severe sepsis or septic shock: a) ≥ 2 systemic inflammatory response syndrome criteria, b) suspected (based on attending physician) or confirmed systemic infection, and c) ≥ 2 or more organ system dysfunctions (severe sepsis) or cardiovascular dysfunction (septic shock).
* An indwelling arterial catheter.
* Parental/guardian permission (informed consent).
* The patient and parent/guardian are fluent in English.

Exclusion Criteria:

* History of neurologic disorder including (hypoxic ischemic injury, traumatic brain injury, epileptic encephalopathy, neurodevelopmental, neurometabolic or neurogenetic conditions, and structural brain anomalies).
* History of cancer or undergoing treatment for cancer.
* Meningitis or encephalitis as source of sepsis.
* Congenital heart disease.
* History of cardiac arrest.
* History of extracorporeal membrane oxygenation (ECMO) cannulation.
* Patients with contraindications to MR scanning.
* Pregnant or lactating females.
* Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.
* Previous enrollment in this study.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children admitted to the pediatric intensive care unit (PICU) at the Children's Hospital of Philadelphia (CHOP) with severe sepsis from an extracranial source and have no history of a preexisting underlying a neurologic disorder.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
MRI | 2-10 days
  Detection of signal abnormality on the patient's brain MRI scan.

SECONDARY OUTCOMES:
CAR | Daily for 10 days
  Trends in functionality of CAR over the first 10 days of severe sepsis. Identification of the optimal blood pressure range where CAR is most functional.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Kirschen, MD, PhD, Principal Investigator — CHOP
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No